CLINICAL TRIAL: NCT01604148
Title: Retrospective Review of a Comprehensive Case Database of HoLEP (Holmium Laser Enucleation of Prostate) Procedure Performed by a Single Surgeon
Brief Title: Retrospective Review a Comprehensive Case Database of HoLEP Procedure Performed by a Single Surgeon
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-06-082
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: Holmium Laser Enucleation of Prostate
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HoLEP group: Holmium Laser Enucleation of Prostate Group

SUMMARY:
Persistent detrusor overactivity (DO) after transurethral prostatectomy results in symptomatic failure in more than one third of the patients. Storage symptoms are major complaints in the early postoperative period after Holmium Laser Enucleation of the Prostate (HoLEP). To investigate the effect of DO in the patients with Benign Prostatic Obstruction (BPO), the investigators evaluated the changes in the storage symptoms following HoLEP in conjunction with the prescription of the anticholinergic drugs.

DETAILED DESCRIPTION:
Eighty men with urodynamically proven BPO underwent HoLEP at our hospital. All patients were evaluated preoperatively with International Prostate Symptom Score (IPSS), International Continence Society male questionnaire short form (ICS-SF), 3-day frequency - volume charts (FVC), transrectal ultrasonography, and uroflowmetry with postvoid residual urine volume. The patients were divided into two groups; BPO without DO (Non-DO group) and BPO with DO (DO group). We assessed the patients postoperatively at 2 weeks, 1, 3 and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* 50 yrs or greater
* International prostatic symptom score >= 12
* Bladder outlet obstruction confirmed by pressure-flow study (BOOI > 20)

Exclusion Criteria:

* Patients with urologic malignancies such as prostate cancer and bladder cancer
* Patients underwent urethral, prostate surgery
* Patients with urethral stricture or bladder diverticulum or bladder neck contracture

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent Holmium Laser Enucleation of the Prostate by a single surgeon
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea